CLINICAL TRIAL: NCT04204668
Title: A Randomized Trial Comparing Surgical Treatments for Neuroma Pain in Amputees
Brief Title: Surgical Treatments for Neuroma Pain in Amputees
Acronym: STOCAP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Johns Hopkins University (Other)
Collaborators: The Plastic Surgery Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00235936
Record Dates: First submitted 2019-12-17; First posted 2019-12-19 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Pain, Neuropathic; Amputation Neuroma; Phantom Limb Pain
MeSH Terms: conditions — Neuralgia; Phantom Limb

STUDY DESIGN:
Intervention Model Description: Three arm, randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Targeted Muscle Reinnervation (TMR) (Active Comparator): In this operation, the surgeon will make a skin incision and carefully identify nerves that were likely to have been injured during the amputation surgery. These nerves are then "cleaned up" to be rerouted and connected to smaller nerves that control individual muscles. The connection to nerves that run into muscles is thought to be helpful in directing the nerve healing process and reducing the risk of developing pain in the future. This operation takes 2 - 4 hours and occurs in the hospital. Follow up requires six to seven clinic visits with the surgeon over the course of one year, at which time standard questionnaires will be used to assess pain.
  Interventions: Procedure: TMR
- Regenerative peripheral nerve interface (RPNI) (Active Comparator): In this operation, the surgeon will make a skin incision and carefully identify nerves that were likely to have been injured during the amputation surgery. The nerves are then "cleaned up" to enhance the possibility of healthy healing. Then the surgeon takes a small sample from a muscle (usually one close by to the nerves that are being operated on but sometimes through a second incision in the arm or leg, depending on the exact medical situation) and form something called a "muscle graft". The muscle graft is used to wrap the cleaned ends of the nerves mentioned above. This is thought to be helpful in directing the nerve healing process and reducing the risk of developing pain in the future. This operation takes 1 - 3 hours and occurs in the hospital. Follow up requires six to seven clinic visits with the surgeon over the course of one year, at which time standard questionnaires will be used to assess pain.
  Interventions: Procedure: RPNI
- Vascularized, denervated muscle target (VDMT ) (Active Comparator): In this operation, the surgeon will make a skin incision and carefully identify nerves that were likely to have been injured during the amputation surgery. The nerves are then "cleaned up" to enhance the possibility of healthy healing. The surgeon will then identify a local muscle along with a small artery and vein that supply blood to part of the muscle. A small sample of muscle, still attached to the artery and vein, is then created. The nearby nerves are then nestled into this segment of muscle that is still connected to the artery and vein. This is thought to be helpful in directing the nerve healing process and reducing the risk of developing pain in the future. This operation takes 2 - 4 hours and occurs in the hospital. Follow up requires six to seven clinic visits with the surgeon over the course of one year, at which time standard questionnaires will be used to assess pain.
  Interventions: Procedure: VDMT

INTERVENTIONS:
Procedure: TMR — Surgical procedure to connect injured proximal nerve stumps to motor nerve branches directly innervating a muscle
  Arms: Targeted Muscle Reinnervation (TMR)
Procedure: RPNI — Surgical procedure to wrap the ends of injured nerves in small muscle grafts
  Arms: Regenerative peripheral nerve interface (RPNI)
Procedure: VDMT — Surgical procedure that creates a small muscle graft that is both denervated and vascularized, which will then receive the damaged nerve ending
  Arms: Vascularized, denervated muscle target (VDMT )

SUMMARY:
Amputees often suffer from relentless pain and disability resulting from symptomatic neuromas within the amputation stumps. When conservative measures fail to address these symptoms, two contemporary surgical approaches to treat symptomatic neuromas have become the most popular. Targeted muscle reinnervation (TMR) is a procedure which involves transferring the injured proximal nerve stump into a terminal nerve branch entering muscle, such that the axons from the proximal nerve stump will regenerate into the muscle and thereby prevent neuroma recurrence. Regenerative peripheral nerve interfaces (RPNIs) are muscle grafts placed on the proximal nerve stumps that serve as targets for the regenerating axons from the proximal nerve stumps.

While TMR and RPNIs have demonstrated promise for the treatment of symptomatic neuromas, prospective comparative data comparing outcomes with these two approaches is lacking.

The investigators have recently developed a novel approach to treat symptomatic neuromas that provides vascularized, denervated muscle targets (VDMTs) for the axons regenerating from the severed proximal nerve stump to reinnervate. This is accomplished by islandizing a segment of muscle on its blood supply and ensuring complete denervation prior to implanting the neighboring transected nerve stump into this muscle. VDMTs offer theoretical benefits in comparison to RPNIs and TMR that the investigators also aim to test in the proposed study.

The investigators' objective is to enroll amputees with symptomatic neuromas into a prospective study in which amputees will be randomized to undergo TMR, RPNI, or VDMT and subsequently monitored for pain and disability for 1-year post-operatively. The investigators' specific aims are as follows: 1) Test the hypothesis that VDMTs are more effective than TMR and RPNIs with regards to treating pain and disability associated with symptomatic neuromas; 2) Provide the first level one, prospective data directly comparing the efficacy of TMR and RPNIs.

DETAILED DESCRIPTION:
Extremity amputations are common operations both in the United States and other areas of the world. It is estimated that there are nearly 2 million adults living in the United States alone. Etiologies for extremity amputation are diverse but the most common indications include complications of type 2 diabetes, non-diabetic peripheral vascular disease, trauma, and oncologic conditions. Given the increasing prevalence of several of these pathologies, conservative estimates suggest that the population of people living with an amputated limb will likely double within the next several decades.

Patients who undergo limb amputation are at significant risk of developing chronic neuropathic pain as a result of symptomatic neuroma formation, due in large part to the abundance of sizeable nerves within the extremities that are necessarily transected as part of the procedure. There are two distinct forms of pain experienced by patients who have undergone major extremity amputations. Residual limb pain is the more straightforward form of post-amputation pain attributable to neuroma formation within the amputation stump. Following peripheral nerve transection, axons regenerating from the proximal stump tend to form aggregates of disorganized neural growth called neuromas. Some neuromas will produce severe, intractable pain causing significant impairment in prosthetic fit and function, activities of daily living, and quality of life. Some estimates place the prevalence of residual limb pain attributable to neuroma formation as high as 75%. The other form of pain is known as phantom limb pain. While the underpinnings of phantom limb pain are the subject of ongoing debate, it is thought by many to arise from chronic stimulation of the cerebral cortex with painful inputs from peripheral neuromas, leading to unpredictable and poorly characterized reorganization of the cortex. Informed estimates of phantom limb pain prevalence as high as 85% have been reported. Successful prevention and treatment of symptomatic neuromas in the setting of limb amputation is therefore of paramount importance given the central role in the pathogenesis of chronic post-amputation limb pain encompassing both residual limb pain and phantom limb pain.

Treatment options for chronic post amputation pain caused by symptomatic neuromas are diverse. Medical options for both phantom limb pain and residual limb pain have been met with limited success. Despite the widespread use, the utility of neuromodulating medications, such as gabapentin, has been called into question by recent large scale meta-analyses that failed to demonstrate meaningful improvements. Neurotoxins, such as botulinum toxin, have also been studied and found to offer limited, if any, pain resolution.

One of the most commonly used surgical approaches to treat and prevent symptomatic neuromas involves burying the proximal nerve stump into nearby muscle. There is a widely-held misconception that burying a proximal nerve stump into muscle will prevent a neuroma from forming. However, elegant animal studies have proven that regeneration of a neuroma is virtually guaranteed because innervated muscle will not accept additional innervation from regenerating neurons.

In the past decade, two other surgical treatments for chronic post-amputation limb pain have come into vogue. Targeted muscle reinnervation (TMR) was initially pioneered as a means of providing intuitive control of advanced prostheses and only later observed to reduce neuroma pain. TMR involves transferring the proximal nerve stump of the injured nerve into a nearby distal motor branch. Early results are promising. A recently published randomized, controlled trial demonstrated the superiority of the TMR approach over the 'bury in muscle' approach, so much so that the trial concluded prematurely due to the superiority of the TMR compared to the historical technique.

The other recently developed and widely popularized option for surgical treatment of chronic post-amputation limb pain involves creation of a regenerative peripheral nerve interface (RPNI). Similar to TMR, the RPNI was initially conceived as a method to provide an interface with an advanced neuroprosthetic prior to being employed as a treatment strategy for neuromas. RPNIs are muscle grafts that are coapted to the ends of severed proximal nerve stumps. This technique has gained popularity because of its technical simplicity and promising early clinical data. In contrast to the 'bury in muscle' approach, RPNIs are denervated at the time of harvest and have been shown to accept reinnervation via direct neurotization from the proximal nerve stump.

To address possible limitations of the strategies described above, the investigators propose using muscle targets similar to RPNIs but maintaining vascularity - a vascularized, denervated muscle target (VDMT). This is accomplished by raising a portion of muscle on a vascular leash in proximity to the transected nerve. Perforating branches from larger blood vessels that perfuse adjacent muscle can be found in abundance throughout the extremities. Any nerves traveling with the vascular leashes will be divided to ensure complete denervation of the muscle. Therefore, VDMTs will be receptive to reinnervation from the implanted proximal nerve stump, maintain vascularity such that the VDMTs can be large enough to supply an abundance of sensory receptors (spindle cells, Golgi apparati, etc) to accept regenerating axons, and avoid the use of a nerve coaptation. In short, the VDMT offers possible enhancements to the surgical techniques currently in use.

In terms of surgical outcomes, there is a robust body of data surrounding the TMR and RPNI operations, with some more recent reports providing pre- and post-operative pain scores for the individual operations. With the exception of one study that prospectively compared TMR to the historical gold standard of neuroma excision and implantation into surrounding tissue, there is a startling lack of prospective data on pain outcomes. Furthermore, the investigators are not aware of prospective, head-to-head comparative data for RPNI vs TMR. Robust, prospective, comparative data is now needed to validate the VDMT approach and assess its efficacy in comparison to the other established techniques.

It is of prime importance to surgeons who perform extremity amputations (eg orthopedic surgeons, vascular surgeons, trauma surgeons, plastic surgeons, and podiatrists) as well as those who perform salvage procedures for post-amputation extremity pain to understand the potential of these operations in treating this pain. Physicians are still lacking evidence-based treatment guidelines. With the generation of this data, surgeons and patients can make more informed decisions about which operative intervention provides the highest likelihood of durable, significant pain relief.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients presenting with > 6 months of intractable post-amputation limb pain with no history of previous surgical intervention for pain treatment.
* Patient is able to sign informed consent and able to participate in all testing associated with this clinical investigation
* Women of childbearing potential who have a negative pregnancy test

Exclusion Criteria:

* Age < 18 years old
* Patient unable to sign informed consent
* Patient participating in another investigational device, surgical technique, or pharmacological study
* Prisoner or patient from vulnerable populations as defined in 45 Code of Federal Regulations (CFR) 46.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
Worst reported residual limb pain score on a numerical scale | One year post-operatively
  Pain score will be assessed using the numerical pain score (0-10) with 0 representing no pain and 10 representing the worst pain.
Worst reported phantom limb pain score on a numerical scale | One year post-operatively
  Pain score will be assessed using the numerical pain score (0-10) with 0 representing no pain and 10 representing the worst pain.

CONTACTS AND LOCATIONS:
Overall Officials: Sami Tuffaha, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No